CLINICAL TRIAL: NCT06725706
Title: Beta Amyloid PET/CT in Various Aβ-Related Disease
Status: Recruiting | Type: Observational
Sponsor: Tianjin Medical University (Other)
Collaborators: Tianjin Medical University General Hospital (Other)
Responsible Party: Principal Investigator, Shaobo Yao, PhD, Prof., Tianjin Medical University
Other Study IDs: TJMUGH-07
Record Dates: First submitted 2024-12-05; First posted 2024-12-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-06

CONDITIONS: Amyloid; Beta-Amyloid; Neurodegenerative Diseases
Keywords: PET/CT; MRI; Beta-Amyloid
MeSH Terms: conditions — Alzheimer Disease; Plaque, Amyloid; Neurodegenerative Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Group Assignment: Each subject receive a single intravenous injection of 18F-92/AV45, 11C-PIB and undergo PET/CT or MRI imaging within the specificed time.
  Interventions: Diagnostic Test: 18F-92/AV45, 11C-PIB

INTERVENTIONS:
Diagnostic Test: 18F-92/AV45, 11C-PIB — Each subject receive a single intravenous injection of 18F-92/AV45, 11C-PIB and undergo PET/CT or MRI imaging within the specificed time.

SUMMARY:
To evaluate the potential usefulness of 18F-92/AV45, 11C-PIB positron emission tomography/computed tomography (PET/CT) for the diagnosis of primary and metastatic lesions in various Tau-related disease patients.

DETAILED DESCRIPTION:
Subjects with various Tau-related disease patients underwent 18F-92/AV45, 11C-PIB PET/CT either for an initial assessment or for recurrence detection. Lesions uptake was quantified by the maximum standard uptake value (SUVmax). The sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV) and accuracy of 18F-92/AV45, 11C-PIB PET/CT were calculated.

ELIGIBILITY:
Inclusion Criteria:

- (i) adult patients (aged 18 years or order); (ii) patients with suspected or new diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report); (iii) patients who had scheduled Aβ PET/CT scan; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

- (i) patients with non-malignant lesions; (ii) patients with pregnancy; (iii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: (i) adult patients (aged 18 years or order); (ii) patients with suspected or new diagnosed or previously treated malignant tumors (supporting evidence may include MRI, CT, tumor markers and pathology report); (iii) patients who had scheduled Aβ PET/CT scan; (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2012-09-01 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value (SUV) | 30 days
  Standardized uptake value (SUV) of 18F-92/AV45, 11C-PIB for each target lesion of subject or suspected primary tumor or/and metastasis.

SECONDARY OUTCOMES:
Diagnostic efficacy | 30 days
  The sensitivity, specificity and accuracy of Aβ PET/CT were calculated.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Chinese PLA General Hospital,, Beijing, Beijing Municipality
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Li Y, Pan M, Yu H, Zhang Q, Chang Y, Zhao H, Wang J, Wang X, Dai J, Yu L, Chen D, Zhang J, Yan XX, Yao S, Cui M. Preclinical and preliminary clinical evaluation of [18F]Florbetazine for non-invasive PET detection of cardiac amyloidosis. Eur J Nucl Med Mol Imaging. 2026 Jan 10. doi: 10.1007/s00259-025-07719-9. Online ahead of print. PMID 41518400